CLINICAL TRIAL: NCT06955702
Title: Effect of Cryotherapy in the Prevention of Alopecia in Eyebrows and Eyelashes in Breast Cancer Patients Treated With Anthracyclines and Taxanes
Brief Title: Effect of Cryotherapy in the Prevention of Madarosis Produced by Chemotherapy in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Marta González Fernández-Conde, PhD, Nursing Professor Ávila School of Nursing (affiliated to University of Salamanca), University of Salamanca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PC_TCUE23-24_033
Record Dates: First submitted 2025-03-26; First posted 2025-05-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Neoplasms; Alopecia; Madarosis; Eyebrow Diseases; Eyelash Diseases; Anthracyclines; Taxoids; Side Effects
Keywords: Chemotherapy-induced alopecia; Madarosis; Eyebrow preservation; Taxane-induced alopecia; Anthracycline-induced alopecia; Cryotherapy; Supportive care in oncology; Quality of life; Scalp cooling; Patient-reported outcomes
MeSH Terms: conditions — Breast Neoplasms; Alopecia | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Quasi-experimental parallel design comparing cryotherapy vs. standard care in two separate patient groups.
Masking Description: Due to the visible nature of cryotherapy, blinding of participants, providers, or assessors was not feasible. Photogrammetric analysis was automated (AI-based) to minimize bias in outcome measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryotherapy on Eyebrows + Chemotherapy (Anthracyclines and Taxanes) (Experimental): Cryotherapy is administered via thermally regulated cold eye masks (-10°C ± 2°C) positioned over the supraorbital region, with application commencing 15 minutes pre-chemotherapy and continuing through the infusion period plus 20 minutes post-administration. Chemotherapy includes anthracyclines (doxorubicin/epirubicin) and/or taxanes (paclitaxel/docetaxel) per standard protocols.
  Interventions: Device: cryotherapy for chemotherapy-induced madarosis
- Standard chemotherapy (no cryotherapy) (No Intervention): Patients receive anthracycline/taxane-based chemotherapy per institutional protocols without application of cold eye masks or any cryotherapy intervention. All other supportive care measures match the experimental group.

INTERVENTIONS:
Device: cryotherapy for chemotherapy-induced madarosis — Application of temperature-controlled cold devices (-4°C to -7°C) to the supraorbital area (up to 3 cm above the eyelid margin), administered 15 minutes before chemotherapy infusion and maintained for 20 minutes post-infusion.
  Arms: Cryotherapy on Eyebrows + Chemotherapy (Anthracyclines and Taxanes)

SUMMARY:
Chemotherapy-induced alopecia (CIA) significantly compromises body image in breast cancer patients, particularly when involving eyebrow and eyelash loss (madarosis). While scalp cooling devices are routinely employed to prevent scalp alopecia, no standardized interventions exist for madarosis prevention. This quasi-experimental study assesses the efficacy of targeted eyebrow cryotherapy in reducing anthracycline- and taxane-induced madarosis.

The trial will enroll patients from two tertiary hospitals in Salamanca (intervention arm: cryotherapy) and a control cohort from Santander. Cryotherapy will be administered (-4°C to -7°C) 15 minutes pre-chemotherapy infusion and maintained for 20 minutes post-infusion. Primary outcomes include hair retention quantified through photogrammetric analysis (TIDOP Research Group) at four timepoints: baseline, mid-treatment, chemotherapy completion, and 1-month follow-up. Secondary endpoints evaluate quality of life (QLQ-C30 validated scales) and cryotherapy-related adverse events (CTCAE v5.0 criteria).

This investigation aims to establish the first evidence-based protocol for madarosis prevention and develop a novel alopecia classification scale, addressing a critical gap in supportive oncology care

DETAILED DESCRIPTION:
Background: Chemotherapy-induced alopecia (CIA) is one of the most distressing adverse effects for breast cancer patients, particularly when involving eyebrow and eyelash loss (madarosis). While scalp cryotherapy has demonstrated efficacy in reducing CIA, no standardized protocols exist for preventing madarosis. Preliminary studies suggest localized cryotherapy may mitigate this effect but robust evidence is lacking.

Objectives: The primary objective is to evaluate the efficacy of supraorbital cryotherapy in preventing anthracycline- or taxane-induced madarosis in breast cancer patients. Secondary objectives include: (1) Quantifying chemotherapy-induced alopecia of eyebrows (madarosis) and eyelashes (milphosis) in control groups, (2) developing a novel alopecia classification scale for eyebrows and eyelashes (currently nonexistent), (3) assessing quality-of-life impact using validated questionnaires "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-BR23 (EORTC QLQ-BR23)" and, and Eyelash Satisfaction Questionnaire (ESQ). (4) monitoring cryotherapy-related adverse events (e.g., headache, localized pain).

Methodology: This non-randomized, quasi-experimental multicenter trial will be conducted at hospitals in Salamanca and Santander. The study population will comprise 120 breast cancer patients receiving anthracycline/taxane-based chemotherapy (sample size may be adjusted based on recruitment). Inclusion criteria: women >18 years old with recent diagnosis and no prior treatments. The intervention group will receive supraorbital cryotherapy using temperature-controlled devices (-4°C to -7°C) applied 15 minutes before chemotherapy infusion and maintained for 20 minutes post-infusion.

Outcome Measures: Primary outcomes will be assessed via:

* Photogrammetric analysis (TIDOP Research Group) at four timepoints: baseline, mid-treatment, end-of-treatment, and 1-month follow-up. Hair retention will be quantified using automated AI algorithms (DAM-Net).
* Patient-reported outcomes using the EORTC QLQ-BR23 and ESQ questionnaires.
* Adverse event monitoring through ad hoc surveys. Statistical Analysis: Data will be analyzed using ANOVA and Mann-Whitney tests for intergroup comparisons, Pearson/Spearman correlations for continuous variables, and linear regression to identify predictive factors.

Ethics: The study has been approved by the Ethics Committees of Salamanca Health Area (Ref: 2023 09 1427) and Hospital Universitario Marqués de Valdecilla (Cantabria, Spain)" (Ref: 2024.459). All participants will provide written informed consent in accordance with the Helsinki Declaration and "General Data Protection Regulation (GDPR)".

Limitations: Current evidence on madarosis/milphosis is limited, and no validated scales exist for grading eyebrow/eyelash alopecia.

Innovations: This study introduces: (1) the first classification scale for chemotherapy-induced madarosis, (2) evidence for cryotherapy as a preventive intervention, and (3) an objective AI-powered photogrammetry methodology.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged ≥18 years
* Newly diagnosed breast cancer (any stage)
* Scheduled to receive anthracycline- and/or taxane-based chemotherapy as first-line systemic treatment
* No prior history of antineoplastic treatment
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients with recurrent disease who have received prior hormone therapy, chemotherapy, and/or immunotherapy
* Presence of alopecia prior to the initiation of cancer treatment
* History of cerebral radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is predominant in women (>99% of cases).
Enrollment: 120 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Eyebrow hair preservation rate | From baseline to 1 month post-chemotherapy completion
  Proportion of patients with ≤50% eyebrow hair loss (Grade 0-2 on CTCAE v5.0 adapted scale) at end of treatment, assessed via AI-based photogrammetry (TIDOP Group)

SECONDARY OUTCOMES:
Eyelash hair preservation rate | From baseline to 1 month post-chemotherapy completion
  Proportion of patients with ≤50% eyelash hair loss (Grade 0-2 on CTCAE v5.0 adapted
Control group madarosis incidence | From baseline to 1 month post-chemotherapy completion
  Absolute reduction in eyebrow hair count (number of hairs lost) from baseline to end-of-treatment, measured via AI-based photogrammetry (DAM-Net)
Change in Body Image Score Measured by EORTC QLQ-BR23 | From baseline to 1 month post-chemotherapy completion
  Mean change in body image subscale score (Items 9-12) from baseline to 1-month post-chemotherapy. Items assess physical attractiveness, femininity, and body dissatisfaction using a 4-point Likert scale (1='Not at all' to 4='Very much'). Raw scores are linearly transformed to a 0-100 scale following EORTC guidelines, where higher scores indicate worse body image perception."*
  Measure: *EORTC QLQ-BR23 (23-item breast cancer-specific module)*
Change in Eyelash Satisfaction measured by Eyelash Satisfaction Questionnaire (ESQ) | From baseline to 1 month post-chemotherapy completion
  Measure: Eyelash Satisfaction Questionnaire (ESQ)
  Description:
  Change in eyelash-related satisfaction assessed through three validated domains of the 23-item ESQ:
  * LFOS (Length, Fullness, Overall Satisfaction): 6 items (Q1-Q6) scored 1-5. Raw sum range: 3-15. Lower scores = Better satisfaction
  * CAP (Confidence, Attractiveness, Professionalism): 7 items (Q16-Q19, Q21-Q23) scored 1-5. Raw sum range: 3-15. Lower scores = Better self-perception
  * DR (Daily Routine): 4 items (Q12-Q15) scored 1-5. Raw sum range: 3-15. Higher scores = Better daily adaptation All items use 5-point Likert scales (1='Very dissatisfied' to 5='Very satisfied'). Scores analyzed as untransformed raw sums per domain."
Cryotherapy-related adverse events | From baseline through chemotherapy completion (approximately 20 to 24 weeks)
  Proportion of patients reporting side effects assessed via a non-validated *ad hoc* questionnaire (Not at all, a little, quite a bit, very much) developed specifically for this study due to lack of validated tools in the literature
Proposal of a new madarosis classification scale | Baseline, after cycles (anthracyclines:4; paclitaxel:8/12*; docetaxel:4/6*), 1mo post-treatment. *if n≥30. Duration: ~1 year
  Development of an automated madarosis grading system through:
  1. Standardized dual-camera imaging: Paired Canon EOS700D (60mm lenses, 1.5m, auto-mode) capturing eyebrow/eyelash regions.
  2. Iterative AI pipeline (Python-based):
     * Phase 1: Temporal alignment via anthropometric landmarks. Deep Learning refinement
     * Phase 2: Pixel-wise hair detection (DAM-Net-class models)
     * Phase 3: Density change analysis
  3. Validation: Against untreated control images Covers most alopecia-inducing drugs in breast cancer (anthracyclines/taxanes). Baseline, post-cycles (anthra:4; pacli:8; docet:4), 1mo post-tx. Additional assessments if n≥30: paclitaxel (12 cycles), docetaxel (6 cycles).
  Open-source release planned.

CONTACTS AND LOCATIONS:
Overall Officials: Marta González Fernández-Conde, Principal Investigator — Universidad Salamanca
Locations (2):
- Spain (2):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Salamanca